CLINICAL TRIAL: NCT00174785
Title: A Placebo-controlled,Double-blind,Parallel Arm Trial to Assess the Efficacy of Dronedarone 400mg Bid for the Prevention of Cardiovascular Hospitalization or Death From Any Cause in Patients With Atrial Fibrillation/Atrial Flutter (AF/AFL)
Brief Title: A Trial With Dronedarone to Prevent Hospitalization or Death in Patients With Atrial Fibrillation
Acronym: ATHENA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: International Clinical Development - Study Director, sanofi-aventis
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: EFC5555
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Results first posted 2009-12-23 (Estimated); Last update posted 2010-01-12 (Estimated); Status verified 2010-01

CONDITIONS: Atrial Fibrillation; Atrial Flutter
Keywords: Mortality, Hospitalization
MeSH Terms: conditions — Atrial Fibrillation; Atrial Flutter | interventions — Dronedarone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dronedarone 400mg bid (Experimental): Dronedarone 400mg tablets twice daily (bid)
  Interventions: Drug: dronedarone (SR33589)
- Placebo (Placebo Comparator): matching placebo tablets
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: dronedarone (SR33589) — oral administration (tablets)
  Other Names: Multaq®
  Arms: Dronedarone 400mg bid
Drug: placebo — oral administration (tablets)
  Arms: Placebo

SUMMARY:
To assess the efficacy of dronedarone in preventing cardiovascular hospitalization or death from any cause in a population of high-risk patients with atrial fibrillation/atrial flutter (AF/AFL).

To assess that dronedarone is well tolerated in this population.

DETAILED DESCRIPTION:
This is a prospective, multinational, double-blind, randomized, multi-center, placebo-controlled, parallel-group trial evaluating the effects of dronedarone versus placebo (ratio 1:1) over a minimum treatment duration of 12 months and a mean follow-up duration of 1.75 years (in AF/AFL patients). Patients can be included in the study while in atrial fibrillation/flutter or in sinus rhythm if conversion has occurred either spontaneously or following a procedure such as electrical cardioversion (or overdrive pacing) or administration of an antiarrhythmic drug.After randomization all patients will be followed until the common study end date; the last patient included in the study will be followed for 1 year. Visits will be at baseline, after 7 days, after 14 days, after one month, after three months and then every three months until end of the study. At each visit patients will be asked for the occurrence of hospitalizations or other events since the last visit. The study will be monitored by an independent Data Monitoring Committee (DMC) for safety, tolerability and efficacy.

ELIGIBILITY:
Inclusion Criteria:

* 1. Patients aged 75 years or older (70 years before protocol amendment 1), or patients aged at least 70 years (any age before protocol amendment 1) with one or more of the following risk factors at baseline:

  * Hypertension (taking antihypertensive drugs of at least two different classes)
  * Diabetes
  * Prior cerebrovascular accident (stroke or transient ischemic attack) or systemic embolism
  * Left atrium diameter greater than or equal to 50 mm by echocardiography
  * Left ventricular ejection fraction less than 0.40 by 2D-echocardiography (two-dimensional echocardiography)
* 2. Availability of one electrocardiogram (ECG) within the last 6 months, showing that the patient was or is in AF/AFL
* 3. Availability of one ECG within the last 6 months, showing that the patient was or is in sinus rhythm

Exclusion Criteria:

General criteria:

* 1. Refusal or inability to give informed consent to participate in the study
* 2. Any non cardiovascular illness or disorder that could preclude participation or severely limit survival including cancer with metastasis and organ transplantation requiring immune suppression
* 3. Pregnant women (pregnancy test must be negative) or women of childbearing potential not on adequate birth control: only women with a highly effective method of contraception [oral contraception or intra-uterine device (IUD)] or sterile can be randomized.
* 4. Breastfeeding women
* 5. Previous (2 preceding months) or current participation in another clinical trial with an investigational drug (under development) or with an investigational device
* 6. Previous participation in this trial

Criteria Related to a cardiac condition:

* 7. Patients in permanent atrial fibrillation
* 8. Patients in unstable hemodynamic condition such as acute pulmonary edema within 12 hours prior to start of study medication; cardiogenic shock; treatment with intra-venous pressor agents; patients on respirator; congestive heart failure of stage NYHA IV (New York Heart Association classification) within the last 4 weeks; uncorrected, hemodynamically significant primary obstructive valvular disease; hemodynamically significant obstructive cardiomyopathy; a cardiac operation or revascularization procedure within 4 weeks preceding randomization
* 9. Planned major non-cardiac or cardiac surgery or procedures including surgery for valvular heart disease, coronary artery bypass graft (CABG) , percutaneous coronary intervention (PCI) , or on urgent cardiac transplantation list
* 10. Acute myocarditis or constrictive pericarditis
* 11. Bradycardia < 50 bpm and/or PR-interval > 0.28 sec on the last 12-lead ECG
* 12. Significant sinus node disease (documented pause of 3 seconds or more) or 2nd or 3rd degree atrioventricular block (AV-block) unless treated with a pacemaker

Criteria Related to Concomitant Medications:

* 13. Need of a concomitant medication that is prohibited in this trial, including the requirement for Vaughan Williams Class I and III anti-arrhythmic drugs, that would preclude the use of study drug during the planned study period

Criteria Related to Laboratory Abnormalities:

* 14. Plasma potassium < 3.5 mmol/l (as anti-arrhythmic drugs can be arrhythmogenic in patients with hypokalemia, this must be corrected prior to randomization)
* 15. A calculated Glomerular Filtration Rate (GFR) at baseline <10 ml/min using the Cockroft Gault formula

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 4628 (Actual)
Dates: Start 2005-06; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: International Clinical Development, Study Director — Sanofi
Locations (37):
- Sanofi-Aventis Administrative Office, Bridgewater, New Jersey, United States
- Sanofi-Aventis Administrative Office, Buenos Aires, Argentina
- Sanofi-Aventis Administrative Office, New South Wales, Australia
- Sanofi-Aventis Administrative Office, Vienna, Austria
- Sanofi-Aventis Administrative Office, Diegem, Belgium
- Sanofi-Aventis Administrative Office, Laval, Canada
- Sanofi-Aventis Administrative Office, Santiago, Chile
- Sanofi-Aventis Administrative Office, Shangaï, China
- Sanofi-Aventis Administrative Office, Prague, Czechia
- Sanofi-Aventis Administrative Office, Helsinki, Finland
- Sanofi-aventis Administrative Office, Berlin, Germany
- Sanofi-Aventis Administrative Office, Athens, Greece
- Sanofi-Aventis Administrative Office, Causeway Bay, Hong Kong
- Sanofi-Aventis Administrative Office, Budapest, Hungary
- Sanofi-Aventis Administrative Office, Mumbai, India
- Sanofi-Aventis Administrative Office, Netanya, Israel
- Sanofi-Aventis Administrative Office, Milan, Italy
- Sanofi-Aventis Administrative Office, Kuala Lumpur, Malaysia
- Sanofi-Aventis Administrative Office, México, Mexico
- Sanofi-Aventis Administrative Office, Casablanca, Morocco
- Sanofi-Aventis Administrative Office, Gouda, Netherlands
- Sanofi-Aventis Administrative Office, Macquarie Park, New Zealand
- Sanofi-Aventis Administrative Office, Lysaker, Norway
- Sanofi-Aventis Administrative Office, Makati City, Philippines
- Sanofi-Aventis Administrative Office, Warsaw, Poland
- Sanofi-Aventis Administrative Office, Porto Salvo, Portugal
- Sanofi-Aventis Administrative Office, Moscow, Russia
- Sanofi-Aventis Administrative Office, Singapore, Singapore
- Sanofi-Aventis Administrative Office, Midrand, South Africa
- Sanofi-Aventis Administrative Office, Seoul, South Korea
- Sanofi-Aventis Administrative Office, Barcelona, Spain
- Sanofi-Aventis Administrative Office, Bromma, Sweden
- Sanofi-Aventis Administrative Office, Taipei, Taiwan
- Sanofi-Aventis Administrative Office, Bangkok, Thailand
- Sanofi-Aventis Administrative Office, Mégrine, Tunisia
- Sanofi-Aventis Administrative Office, Istanbul, Turkey (Türkiye)
- Sanofi-Aventis Administrative Office, Guildford Surrey, United Kingdom

REFERENCES:
- [Background] Hohnloser SH, Connolly SJ, Crijns HJ, Page RL, Seiz W, Torp-Petersen C. Rationale and design of ATHENA: A placebo-controlled, double-blind, parallel arm Trial to assess the efficacy of dronedarone 400 mg bid for the prevention of cardiovascular Hospitalization or death from any cause in patiENts with Atrial fibrillation/atrial flutter. J Cardiovasc Electrophysiol. 2008 Jan;19(1):69-73. doi: 10.1111/j.1540-8167.2007.01016.x. Epub 2007 Nov 21. PMID 18031520
- [Result] Hohnloser SH, Crijns HJ, van Eickels M, Gaudin C, Page RL, Torp-Pedersen C, Connolly SJ; ATHENA Investigators. Effect of dronedarone on cardiovascular events in atrial fibrillation. N Engl J Med. 2009 Feb 12;360(7):668-78. doi: 10.1056/NEJMoa0803778. PMID 19213680
- [Derived] Kirchhof P, Camm AJ, Crijns HJGM, Piccini JP, Torp-Pedersen C, McKindley DS, Wieloch M, Hohnloser SH. Dronedarone provides effective early rhythm control: post-hoc analysis of the ATHENA trial using EAST-AFNET 4 criteria. Europace. 2025 Mar 28;27(4):euaf080. doi: 10.1093/europace/euaf080. PMID 40295782
- [Derived] Handelsman Y, Bunch TJ, Rodbard HW, Steinberg BA, Thind M, Bigot G, Konigsberg L, Wieloch M, Kowey PR. Impact of dronedarone on patients with atrial fibrillation and diabetes: A sub-analysis of the ATHENA and EURIDIS/ADONIS studies. J Diabetes Complications. 2022 Jul;36(7):108227. doi: 10.1016/j.jdiacomp.2022.108227. Epub 2022 Jun 8. PMID 35717354
- [Derived] Vamos M, Oldgren J, Nam GB, Lip GYH, Calkins H, Zhu J, Ueng KC, Ludwigs U, Wieloch M, Stewart J, Hohnloser SH. Dronedarone vs. placebo in patients with atrial fibrillation or atrial flutter across a range of renal function: a post hoc analysis of the ATHENA trial. Eur Heart J Cardiovasc Pharmacother. 2022 Jun 8;8(4):363-371. doi: 10.1093/ehjcvp/pvab090. PMID 34958366
- [Derived] Akerborg O, Nilsson J, Bascle S, Lindgren P, Reynolds M. Cost-effectiveness of dronedarone in atrial fibrillation: results for Canada, Italy, Sweden, and Switzerland. Clin Ther. 2012 Aug;34(8):1788-802. doi: 10.1016/j.clinthera.2012.06.007. Epub 2012 Jul 6. PMID 22770643
- [Derived] Torp-Pedersen C, Crijns HJ, Gaudin C, Page RL, Connolly SJ, Hohnloser SH; ATHENA Investigators. Impact of dronedarone on hospitalization burden in patients with atrial fibrillation: results from the ATHENA study. Europace. 2011 Aug;13(8):1118-26. doi: 10.1093/europace/eur102. Epub 2011 May 15. PMID 21576129
- [Derived] Page RL, Connolly SJ, Crijns HJ, van Eickels M, Gaudin C, Torp-Pedersen C, Hohnloser SH; ATHENA Investigators. Rhythm- and rate-controlling effects of dronedarone in patients with atrial fibrillation (from the ATHENA trial). Am J Cardiol. 2011 Apr 1;107(7):1019-22. doi: 10.1016/j.amjcard.2010.11.028. Epub 2011 Feb 4. PMID 21296333
- [Derived] Hohnloser SH, Crijns HJ, van Eickels M, Gaudin C, Page RL, Torp-Pedersen C, Connolly SJ; ATHENA Investigators. Dronedarone in patients with congestive heart failure: insights from ATHENA. Eur Heart J. 2010 Jul;31(14):1717-21. doi: 10.1093/eurheartj/ehq113. Epub 2010 Apr 30. PMID 20436046
- See also: Related Info — http://www.sanofi-aventis.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment of patients started on June 29, 2005 and was completed on December 30, 2006. The study was conducted at 551 centers in 37 countries. The common study end date ensuring a minimum planned follow-up of one year was December 30th, 2007.
Groups:
- Dronedarone 400mg Bid: dronedarone tablets 400mg twice daily
Period: Overall Study
Arm/Group | Dronedarone 400mg Bid | Placebo
Started | 2301 (randomized patients; among them, 10 patients did not receive any study drug in the dronedarone group) | 2327 (randomized patients; among them, 14 patients did not receive any study drug in the placebo group)
Completed | 1605 (completed study drug) | 1611 (completed study drug)
Not Completed | 696 | 716
Not completed — Adverse Event | 293 | 191
Not completed — Protocol Violation | 14 | 14
Not completed — Withdrawal by Subject | 173 | 175
Not completed — Atrial Fibrillation/Flutter recurrence | 110 | 167
Not completed — Prohibited antiarrhythmic medication | 39 | 88
Not completed — Other prohibited medication | 5 | 3
Not completed — Family request | 6 | 8
Not completed — Not pre-specified/Not coded | 56 | 70

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dronedarone 400mg Bid | Placebo | Total
Number analyzed (Participants) | 2301 | 2327 | 4628
Age, Customized [Number; unit: participants]
  18 to < 65 years | 431 | 442 | 873
  65 to < 75 years | 923 | 907 | 1830
  >= 75 years | 947 | 978 | 1925
Age Continuous [Mean (Standard Deviation); unit: years] | 71.6 (8.9) | 71.7 (9.0) | 71.6 (9.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1131 | 1038 | 2169
  Male | 1170 | 1289 | 2459

OUTCOME MEASURES:

1. Primary Outcome: First Hospitalization for Cardiovascular Reason or Death From Any Cause
Description: The primary event is the first hospitalization for cardiovascular reason or death from any cause, whichever is earlier, as assessed by the investigator. The primary efficacy analysis is performed on the time from randomization to this primary event. The Measured Values table below presents the numbers of patients with the event at the end of the study period.
Time Frame: minimum follow-up duration: 1 year ; maximum: 2.5 years
Population: All efficacy analyses were performed on the "all randomized patients" population including all patients randomized irrespective of whether the patient actually received any drug or complied with the study protocol.
Measure: Number; unit: participants
Arm/Group | Dronedarone 400mg Bid | Placebo
Number analyzed (Participants) | 2301 | 2327
participants | 734 | 917
Statistical Analysis 1: Comparison: Dronedarone 400mg Bid vs Placebo; Test type: Superiority or Other; p < 0.0001, Log Rank — Cumulative incidence functions in each treatment group were calculated using non-parametric Kaplan-Meier estimates. Median time-to-event was not reached in any group. The primary comparison was performed at the 5% level using a 2-sided Log rank test; Hazard Ratio (HR) = 0.76, 95% CI [0.69 to 0.84] — The hazard ratio was estimated by a Cox's proportional hazard model with treatment arm factor. It represents the relative hazard of first hospitalization for cardiovascular reason or death for the dronedarone group compared with the placebo group

2. Secondary Outcome: Death From Any Cause
Description: The considered event is death from any cause. The analysis is performed on the time from randomization to this event. The Measured Values table below presents the numbers of patients with the event at the end of the study period.
Time Frame: minimum follow-up duration: 1 year ; maximum: 2.5 years
Population: "All randomized patients" population
Measure: Number; unit: participants
Arm/Group | Dronedarone 400mg Bid | Placebo
Number analyzed (Participants) | 2301 | 2327
participants | 116 | 139
Statistical Analysis 1: Comparison: Dronedarone 400mg Bid vs Placebo; Test type: Superiority or Other; p = 0.18, Log Rank — Cumulative incidences calculated in each group using non-parametric Kaplan-Meier estimates. Median time-to-event was not reached in any group. Hierarchical procedure applied to secondary efficacy endpoints testing to protect the global type I error; Hazard Ratio (HR) = 0.84, 95% CI [0.66 to 1.08] — The hazard ratio was estimated by a Cox's proportional hazard model with treatment arm factor. It represents the relative hazard of death from any cause for the dronedarone group compared with the placebo group

3. Secondary Outcome: First Hospitalization for Cardiovascular Reason
Description: The considered event is the first hospitalization for cardiovascular reason, as assessed by the Investigator. The analysis is performed on the time from randomization to this event. The Measured Values table below presents the numbers of patients with the event at the end of the study period.
Time Frame: minimum follow-up duration: 1 year ; maximum: 2.5 years
Population: "All randomized patients" population
Measure: Number; unit: participants
Arm/Group | Dronedarone 400mg Bid | Placebo
Number analyzed (Participants) | 2301 | 2327
participants | 675 | 859
Statistical Analysis 1: Comparison: Dronedarone 400mg Bid vs Placebo; Test type: Superiority or Other; p < 0.0001, Log Rank — [p-value comment as in outcome 2, analysis 1]; Hazard Ratio (HR) = 0.74, 95% CI [0.67 to 0.82] — The hazard ratio was estimated by a Cox's proportional hazard model with treatment arm factor. It represents the relative hazard of first hospitalization for cardiovascular reason for the dronedarone group compared with the placebo group

4. Secondary Outcome: Cardiovascular Death
Description: The considered event is cardiovascular death, as assessed by the Investigator. The analysis is performed on the time from randomization to this event. The Measured Values table below presents the numbers of patients with the event at the end of the study period.
Time Frame: minimum follow-up duration: 1 year ; maximum: 2.5 years
Population: "All randomized patients" population
Measure: Number; unit: participants
Arm/Group | Dronedarone 400mg Bid | Placebo
Number analyzed (Participants) | 2301 | 2327
participants | 65 | 94
Statistical Analysis 1: Comparison: Dronedarone 400mg Bid vs Placebo; Test type: Superiority or Other; p = 0.025, Log Rank — [p-value comment as in outcome 2, analysis 1]; Hazard Ratio (HR) = 0.70, 95% CI [0.51 to 0.96] — The hazard ratio was estimated by a Cox's proportional hazard model with treatment arm factor. It represents the relative hazard of cardiovascular death for the dronedarone group compared with the placebo group

5. Other Pre Specified Outcome: Adjudicated Cardiovascular Death
Description: The considered event is cardiovascular death, as assessed by the blinded adjudication of the Steering Committee. The analysis is performed on the time from randomization to this event. The Measured Values table below presents the numbers of patients with the event at the end of the study period.
Time Frame: minimum follow-up duration: 1 year ; maximum: 2.5 years
Population: "All randomized patients" population
Measure: Number; unit: participants
Arm/Group | Dronedarone 400mg Bid | Placebo
Number analyzed (Participants) | 2301 | 2327
participants | 63 | 90
Statistical Analysis 1: Comparison: Dronedarone 400mg Bid vs Placebo; Test type: Superiority or Other; p = 0.03, Log Rank — Cumulative incidences calculated in each group using non-parametric Kaplan-Meier estimates. Median time-to-event was not reached in any group. The comparison was performed at the 5% level using a 2-sided Log rank; Hazard Ratio (HR) = 0.71, 95% CI [0.51 to 0.98] — The hazard ratio was estimated by a Cox's proportional hazard model with treatment arm factor. It represents the relative hazard of adjudicated cardiovascular death for the dronedarone group compared with the placebo group

ADVERSE EVENTS:
Time Frame: In both treatment groups, the median duration of exposure was about 18 months, with a maximum of 30 months.
Description: Reported Events are Treatment-Emergent Adverse Events with an onset date between the first study drug intake and the last study drug intake + 10 days and any pre-treatment adverse event that led to study drug permanent discontinuation.
Arm/Group | Dronedarone 400mg Bid | Placebo
Serious Adverse Events (participants affected / at risk) | 456/2291 | 489/2313
Other Adverse Events (participants affected / at risk) | 1584/2291 | 1527/2313
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dronedarone 400mg Bid (N=2291) | Placebo (N=2313)
Pneumonia (Infections and infestations) | 32 | 45
Urinary tract infection (Infections and infestations) | 6 | 10
Cellulitis (Infections and infestations) | 5 | 7
Gastroenteritis (Infections and infestations) | 5 | 6
Lobar pneumonia (Infections and infestations) | 5 | 6
Diverticulitis (Infections and infestations) | 4 | 4
Bronchitis (Infections and infestations) | 4 | 3
Appendicitis (Infections and infestations) | 4 | 2
Bronchopneumonia (Infections and infestations) | 4 | 2
Sepsis (Infections and infestations) | 3 | 3
Urosepsis (Infections and infestations) | 2 | 4
Pyelonephritis chronic (Infections and infestations) | 2 | 2
Herpes zoster (Infections and infestations) | 2 | 1
Pyelonephritis (Infections and infestations) | 2 | 1
Bronchiectasis (Infections and infestations) | 2 | 0
Mastitis (Infections and infestations) | 2 | 0
Respiratory tract infection viral (Infections and infestations) | 2 | 0
Septic shock (Infections and infestations) | 1 | 4
Upper respiratory tract infection (Infections and infestations) | 1 | 3
Viral infection (Infections and infestations) | 1 | 1
Abscess (Infections and infestations) | 1 | 0
Abscess limb (Infections and infestations) | 1 | 0
Abscess oral (Infections and infestations) | 1 | 0
Acarodermatitis (Infections and infestations) | 1 | 0
Clonorchiasis (Infections and infestations) | 1 | 0
Diarrhoea infectious (Infections and infestations) | 1 | 0
Encephalitis viral (Infections and infestations) | 1 | 0
Epstein-barr virus infection (Infections and infestations) | 1 | 0
Escherichia sepsis (Infections and infestations) | 1 | 0
Gastroenteritis viral (Infections and infestations) | 1 | 0
Hepatitis a (Infections and infestations) | 1 | 0
Infected epidermal cyst (Infections and infestations) | 1 | 0
Infection (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 1 | 0
Localised infection (Infections and infestations) | 1 | 0
Opisthorchiasis (Infections and infestations) | 1 | 0
Orchitis (Infections and infestations) | 1 | 0
Osteomyelitis (Infections and infestations) | 1 | 0
Osteomyelitis chronic (Infections and infestations) | 1 | 0
Pancreatitis viral (Infections and infestations) | 1 | 0
Peritoneal infection (Infections and infestations) | 1 | 0
Pneumonia bacterial (Infections and infestations) | 1 | 0
Pneumonia klebsiella (Infections and infestations) | 1 | 0
Rectal abscess (Infections and infestations) | 1 | 0
Respiratory tract infection (Infections and infestations) | 1 | 0
Skin infection (Infections and infestations) | 1 | 0
Soft tissue infection (Infections and infestations) | 1 | 0
Wound infection bacterial (Infections and infestations) | 1 | 0
Erysipelas (Infections and infestations) | 0 | 4
Device related infection (Infections and infestations) | 0 | 3
Sinusitis (Infections and infestations) | 0 | 3
Clostridium difficile colitis (Infections and infestations) | 0 | 2
Obstructive chronic bronchitis with acute exacerbation (Infections and infestations) | 0 | 2
Postoperative wound infection (Infections and infestations) | 0 | 2
Pyelonephritis acute (Infections and infestations) | 0 | 2
Abdominal abscess (Infections and infestations) | 0 | 1
Bacteraemia (Infections and infestations) | 0 | 1
Bursitis infective (Infections and infestations) | 0 | 1
Diabetic gangrene (Infections and infestations) | 0 | 1
Gastroenteritis salmonella (Infections and infestations) | 0 | 1
Groin infection (Infections and infestations) | 0 | 1
Hiv infection (Infections and infestations) | 0 | 1
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 0 | 1
Labyrinthitis (Infections and infestations) | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 0 | 1
Paronychia (Infections and infestations) | 0 | 1
Peridiverticular abscess (Infections and infestations) | 0 | 1
Peritonsillar abscess (Infections and infestations) | 0 | 1
Pneumonia legionella (Infections and infestations) | 0 | 1
Pneumonia pneumococcal (Infections and infestations) | 0 | 1
Pneumonia staphylococcal (Infections and infestations) | 0 | 1
Post procedural infection (Infections and infestations) | 0 | 1
Pyothorax (Infections and infestations) | 0 | 1
Staphylococcal infection (Infections and infestations) | 0 | 1
Staphylococcal sepsis (Infections and infestations) | 0 | 1
Tinea cruris (Infections and infestations) | 0 | 1
Tracheobronchitis (Infections and infestations) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 6 | 5
Diarrhoea (Gastrointestinal disorders) | 6 | 4
Gastritis (Gastrointestinal disorders) | 5 | 4
Pancreatitis acute (Gastrointestinal disorders) | 4 | 3
Abdominal pain (Gastrointestinal disorders) | 4 | 2
Small intestinal obstruction (Gastrointestinal disorders) | 4 | 1
Inguinal hernia (Gastrointestinal disorders) | 3 | 3
Colonic polyp (Gastrointestinal disorders) | 3 | 1
Pancreatitis (Gastrointestinal disorders) | 3 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 | 3
Abdominal pain upper (Gastrointestinal disorders) | 2 | 2
Nausea (Gastrointestinal disorders) | 2 | 2
Abdominal adhesions (Gastrointestinal disorders) | 2 | 0
Abdominal hernia (Gastrointestinal disorders) | 2 | 0
Abdominal strangulated hernia (Gastrointestinal disorders) | 2 | 0
Constipation (Gastrointestinal disorders) | 2 | 0
Crohn's disease (Gastrointestinal disorders) | 2 | 0
Gastric haemorrhage (Gastrointestinal disorders) | 2 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 2 | 0
Ileus (Gastrointestinal disorders) | 2 | 0
Mallory-weiss syndrome (Gastrointestinal disorders) | 2 | 0
Vomiting (Gastrointestinal disorders) | 2 | 0
Gastric ulcer (Gastrointestinal disorders) | 1 | 3
Intestinal obstruction (Gastrointestinal disorders) | 1 | 3
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 3
Colitis (Gastrointestinal disorders) | 1 | 2
Colitis ischaemic (Gastrointestinal disorders) | 1 | 2
Thrombosis mesenteric vessel (Gastrointestinal disorders) | 1 | 2
Oesophagitis (Gastrointestinal disorders) | 1 | 1
Anal prolapse (Gastrointestinal disorders) | 1 | 0
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 1 | 0
Duodenal ulcer (Gastrointestinal disorders) | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0
Femoral hernia, obstructive (Gastrointestinal disorders) | 1 | 0
Food poisoning (Gastrointestinal disorders) | 1 | 0
Gastritis erosive (Gastrointestinal disorders) | 1 | 0
Gastritis haemorrhagic (Gastrointestinal disorders) | 1 | 0
Gastroduodenitis (Gastrointestinal disorders) | 1 | 0
Ileus paralytic (Gastrointestinal disorders) | 1 | 0
Infrequent bowel movements (Gastrointestinal disorders) | 1 | 0
Intestinal fistula (Gastrointestinal disorders) | 1 | 0
Lumbar hernia (Gastrointestinal disorders) | 1 | 0
Mouth haemorrhage (Gastrointestinal disorders) | 1 | 0
Oesophageal mass (Gastrointestinal disorders) | 1 | 0
Oesophageal spasm (Gastrointestinal disorders) | 1 | 0
Oesophagitis ulcerative (Gastrointestinal disorders) | 1 | 0
Peritonitis (Gastrointestinal disorders) | 1 | 0
Reflux oesophagitis (Gastrointestinal disorders) | 1 | 0
Toothache (Gastrointestinal disorders) | 1 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Appendicitis perforated (Gastrointestinal disorders) | 0 | 2
Diverticulum (Gastrointestinal disorders) | 0 | 2
Dysphagia (Gastrointestinal disorders) | 0 | 2
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 | 2
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 2
Colitis ulcerative (Gastrointestinal disorders) | 0 | 1
Diverticular perforation (Gastrointestinal disorders) | 0 | 1
Diverticulum intestinal (Gastrointestinal disorders) | 0 | 1
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1
Gastric polyps (Gastrointestinal disorders) | 0 | 1
Haematemesis (Gastrointestinal disorders) | 0 | 1
Haematochezia (Gastrointestinal disorders) | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 1
Hiatus hernia, obstructive (Gastrointestinal disorders) | 0 | 1
Intestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Intussusception (Gastrointestinal disorders) | 0 | 1
Irritable bowel syndrome (Gastrointestinal disorders) | 0 | 1
Mesenteric artery thrombosis (Gastrointestinal disorders) | 0 | 1
Mesenteric occlusion (Gastrointestinal disorders) | 0 | 1
Oedematous pancreatitis (Gastrointestinal disorders) | 0 | 1
Peptic ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1
Short-bowel syndrome (Gastrointestinal disorders) | 0 | 1
Umbilical hernia (Gastrointestinal disorders) | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 | 11
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 5
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 5
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 3
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Oesophageal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Renal cell carcinoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 3
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Lung squamous cell carcinoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Prostatic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Hepatic neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Lung adenocarcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Non-small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Benign neoplasm of thyroid gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bladder papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bronchioloalveolar carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Carcinoid tumour pulmonary (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Hepatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Leiomyosarcoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastatic carcinoma of the bladder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Multiple myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Myeloproliferative disorder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Nasal cavity cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Oesophageal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pancreatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Rectal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Thymoma malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Urethral adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Ovarian adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Adrenal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Benign peritoneal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Breast cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Breast cancer stage iii (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Inflammatory carcinoma of the breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Large intestine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lip and/or oral cavity cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Ocular neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Papillary serous endometrial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Pituitary tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Plasmacytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Pleura carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Small cell lung cancer stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Tumour ulceration (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Vulval cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 20 | 20
Hip fracture (Injury, poisoning and procedural complications) | 5 | 2
Road traffic accident (Injury, poisoning and procedural complications) | 3 | 3
Contusion (Injury, poisoning and procedural complications) | 3 | 2
Femoral neck fracture (Injury, poisoning and procedural complications) | 3 | 0
Therapeutic agent toxicity (Injury, poisoning and procedural complications) | 3 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 2 | 2
Accidental overdose (Injury, poisoning and procedural complications) | 2 | 1
Femur fracture (Injury, poisoning and procedural complications) | 2 | 1
Rib fracture (Injury, poisoning and procedural complications) | 2 | 1
Alcohol poisoning (Injury, poisoning and procedural complications) | 2 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 2 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 4
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 3
Traumatic haematoma (Injury, poisoning and procedural complications) | 1 | 3
Brain contusion (Injury, poisoning and procedural complications) | 1 | 2
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 | 1
Post procedural haematoma (Injury, poisoning and procedural complications) | 1 | 1
Post-traumatic pain (Injury, poisoning and procedural complications) | 1 | 1
Pubic rami fracture (Injury, poisoning and procedural complications) | 1 | 1
Skull fracture (Injury, poisoning and procedural complications) | 1 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 1
Traumatic arthritis (Injury, poisoning and procedural complications) | 1 | 1
Acetabulum fracture (Injury, poisoning and procedural complications) | 1 | 0
Anaemia postoperative (Injury, poisoning and procedural complications) | 1 | 0
Anastomotic complication (Injury, poisoning and procedural complications) | 1 | 0
Asbestosis (Injury, poisoning and procedural complications) | 1 | 0
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0
Device failure (Injury, poisoning and procedural complications) | 1 | 0
Foot fracture (Injury, poisoning and procedural complications) | 1 | 0
Head injury (Injury, poisoning and procedural complications) | 1 | 0
Incisional hernia (Injury, poisoning and procedural complications) | 1 | 0
Joint injury (Injury, poisoning and procedural complications) | 1 | 0
Medical device pain (Injury, poisoning and procedural complications) | 1 | 0
Patella fracture (Injury, poisoning and procedural complications) | 1 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Postoperative heterotopic calcification (Injury, poisoning and procedural complications) | 1 | 0
Transfusion reaction (Injury, poisoning and procedural complications) | 1 | 0
Dislocation of joint prosthesis (Injury, poisoning and procedural complications) | 0 | 5
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 3
Arterial injury (Injury, poisoning and procedural complications) | 0 | 1
Concussion (Injury, poisoning and procedural complications) | 0 | 1
Device migration (Injury, poisoning and procedural complications) | 0 | 1
Facial bones fracture (Injury, poisoning and procedural complications) | 0 | 1
Fibula fracture (Injury, poisoning and procedural complications) | 0 | 1
Graft thrombosis (Injury, poisoning and procedural complications) | 0 | 1
Hand fracture (Injury, poisoning and procedural complications) | 0 | 1
Injury (Injury, poisoning and procedural complications) | 0 | 1
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 1
Muscle injury (Injury, poisoning and procedural complications) | 0 | 1
Operative haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 0 | 1
Pelvic fracture (Injury, poisoning and procedural complications) | 0 | 1
Penetrating abdominal trauma (Injury, poisoning and procedural complications) | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 0 | 1
Spinal cord injury cervical (Injury, poisoning and procedural complications) | 0 | 1
Traumatic arthropathy (Injury, poisoning and procedural complications) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 13 | 19
Asthma (Respiratory, thoracic and mediastinal disorders) | 5 | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 4 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 | 4
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Emphysema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal turbinate hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Bronchopneumopathy (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 15 | 21
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 2
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 | 2
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 2 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 5
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 4
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 | 4
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 3
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 2
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 | 1
Arthropathy (Musculoskeletal and connective tissue disorders) | 1 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Dupuytren's contracture (Musculoskeletal and connective tissue disorders) | 1 | 0
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0
Spondylolisthesis acquired (Musculoskeletal and connective tissue disorders) | 1 | 0
Sympathetic posterior cervical syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Intervertebral disc compression (Musculoskeletal and connective tissue disorders) | 0 | 1
Neck mass (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteoporotic fracture (Musculoskeletal and connective tissue disorders) | 0 | 1
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 1
Polyarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 0 | 1
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 1
Spondylolysis (Musculoskeletal and connective tissue disorders) | 0 | 1
Renal failure acute (Renal and urinary disorders) | 14 | 4
Haematuria (Renal and urinary disorders) | 7 | 7
Calculus urinary (Renal and urinary disorders) | 2 | 2
Nephrolithiasis (Renal and urinary disorders) | 2 | 2
Diabetic nephropathy (Renal and urinary disorders) | 2 | 0
Hydronephrosis (Renal and urinary disorders) | 1 | 2
Urinary retention (Renal and urinary disorders) | 1 | 2
Renal colic (Renal and urinary disorders) | 1 | 1
Renal failure (Renal and urinary disorders) | 1 | 1
Renal failure chronic (Renal and urinary disorders) | 1 | 1
Calculus bladder (Renal and urinary disorders) | 1 | 0
Nocturia (Renal and urinary disorders) | 1 | 0
Renal impairment (Renal and urinary disorders) | 1 | 0
Urinary bladder polyp (Renal and urinary disorders) | 1 | 0
Bladder obstruction (Renal and urinary disorders) | 0 | 1
Cystitis haemorrhagic (Renal and urinary disorders) | 0 | 1
Cystitis noninfective (Renal and urinary disorders) | 0 | 1
Stress urinary incontinence (Renal and urinary disorders) | 0 | 1
Urethral stenosis (Renal and urinary disorders) | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 6 | 5
Cholecystitis (Hepatobiliary disorders) | 6 | 4
Cholangitis (Hepatobiliary disorders) | 4 | 0
Cholelithiasis (Hepatobiliary disorders) | 3 | 7
Bile duct stone (Hepatobiliary disorders) | 2 | 1
Biliary colic (Hepatobiliary disorders) | 2 | 0
Cholecystitis chronic (Hepatobiliary disorders) | 1 | 2
Hepatitis toxic (Hepatobiliary disorders) | 1 | 0
Jaundice (Hepatobiliary disorders) | 1 | 0
Hepatic cirrhosis (Hepatobiliary disorders) | 0 | 2
Cholestasis (Hepatobiliary disorders) | 0 | 1
Cytolytic hepatitis (Hepatobiliary disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 4 | 10
Diabetes mellitus (Metabolism and nutrition disorders) | 4 | 3
Hypoglycaemia (Metabolism and nutrition disorders) | 3 | 3
Hyponatraemia (Metabolism and nutrition disorders) | 3 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 3
Gout (Metabolism and nutrition disorders) | 1 | 2
Anorexia (Metabolism and nutrition disorders) | 1 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 1
Fluid overload (Metabolism and nutrition disorders) | 1 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 1 | 0
Vitamin b12 deficiency (Metabolism and nutrition disorders) | 1 | 0
Failure to thrive (Metabolism and nutrition disorders) | 0 | 1
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1
Dizziness (Nervous system disorders) | 3 | 2
Transient ischaemic attack (Nervous system disorders) | 2 | 2
Dementia alzheimer's type (Nervous system disorders) | 2 | 1
Ischaemic stroke (Nervous system disorders) | 2 | 1
Sciatica (Nervous system disorders) | 2 | 1
Syncope (Nervous system disorders) | 1 | 1
Brain mass (Nervous system disorders) | 1 | 0
Cerebrovascular disorder (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 0
Intracranial aneurysm (Nervous system disorders) | 1 | 0
Lumbar radiculopathy (Nervous system disorders) | 1 | 0
Pseudobulbar palsy (Nervous system disorders) | 1 | 0
Spinal claudication (Nervous system disorders) | 1 | 0
Vascular encephalopathy (Nervous system disorders) | 1 | 0
Vertebrobasilar insufficiency (Nervous system disorders) | 1 | 0
Carpal tunnel syndrome (Nervous system disorders) | 0 | 3
Cerebrovascular accident (Nervous system disorders) | 0 | 2
Partial seizures (Nervous system disorders) | 0 | 2
Amyotrophic lateral sclerosis (Nervous system disorders) | 0 | 1
Convulsion (Nervous system disorders) | 0 | 1
Diplegia (Nervous system disorders) | 0 | 1
Epilepsy (Nervous system disorders) | 0 | 1
Facial palsy (Nervous system disorders) | 0 | 1
Guillain-barre syndrome (Nervous system disorders) | 0 | 1
Haemorrhagic stroke (Nervous system disorders) | 0 | 1
Hepatic encephalopathy (Nervous system disorders) | 0 | 1
Loss of consciousness (Nervous system disorders) | 0 | 1
Metabolic encephalopathy (Nervous system disorders) | 0 | 1
Mononeuritis (Nervous system disorders) | 0 | 1
Toxic encephalopathy (Nervous system disorders) | 0 | 1
Blood creatinine increased (Investigations) | 5 | 1
International normalised ratio increased (Investigations) | 4 | 6
Electrocardiogram qt prolonged (Investigations) | 4 | 1
Weight decreased (Investigations) | 1 | 1
Cardioactive drug level increased (Investigations) | 1 | 0
Coagulation test abnormal (Investigations) | 1 | 0
International normalised ratio decreased (Investigations) | 1 | 0
Prothrombin time prolonged (Investigations) | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 1
Blood creatine phosphokinase increased (Investigations) | 0 | 1
Glycosylated haemoglobin increased (Investigations) | 0 | 1
Hepatitis c positive (Investigations) | 0 | 1
Transaminases increased (Investigations) | 0 | 1
Bradycardia (Cardiac disorders) | 2 | 3
Cardiac failure (Cardiac disorders) | 2 | 2
Pericardial effusion (Cardiac disorders) | 2 | 1
Ventricular tachycardia (Cardiac disorders) | 1 | 1
Acute myocardial infarction (Cardiac disorders) | 1 | 0
Angina pectoris (Cardiac disorders) | 1 | 0
Cardiac tamponade (Cardiac disorders) | 1 | 0
Coronary artery disease (Cardiac disorders) | 1 | 0
Pericardial haemorrhage (Cardiac disorders) | 1 | 0
Sinus bradycardia (Cardiac disorders) | 1 | 0
Torsade de pointes (Cardiac disorders) | 1 | 0
Ventricle rupture (Cardiac disorders) | 1 | 0
Ventricular extrasystoles (Cardiac disorders) | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 2
Angina unstable (Cardiac disorders) | 0 | 1
Aortic valve calcification (Cardiac disorders) | 0 | 1
Aortic valve incompetence (Cardiac disorders) | 0 | 1
Atrioventricular block complete (Cardiac disorders) | 0 | 1
Cardiac perforation (Cardiac disorders) | 0 | 1
Right ventricular failure (Cardiac disorders) | 0 | 1
Ventricular flutter (Cardiac disorders) | 0 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 8 | 10
Uterine polyp (Reproductive system and breast disorders) | 1 | 1
Acquired hydrocele (Reproductive system and breast disorders) | 1 | 0
Breast discomfort (Reproductive system and breast disorders) | 1 | 0
Endometrial hyperplasia (Reproductive system and breast disorders) | 1 | 0
Penis disorder (Reproductive system and breast disorders) | 1 | 0
Uterine prolapse (Reproductive system and breast disorders) | 1 | 0
Prostatitis (Reproductive system and breast disorders) | 0 | 3
Vaginal prolapse (Reproductive system and breast disorders) | 0 | 2
Adnexa uteri cyst (Reproductive system and breast disorders) | 0 | 1
Epididymitis (Reproductive system and breast disorders) | 0 | 1
Gynaecomastia (Reproductive system and breast disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 4 | 3
Asthenia (General disorders) | 3 | 3
Pyrexia (General disorders) | 2 | 2
General physical health deterioration (General disorders) | 1 | 2
Drowning (General disorders) | 1 | 0
Oedema (General disorders) | 1 | 0
Oedema peripheral (General disorders) | 1 | 0
Multi-organ failure (General disorders) | 0 | 2
Hernia (General disorders) | 0 | 1
Impaired healing (General disorders) | 0 | 1
Implant site haematoma (General disorders) | 0 | 1
Injection site haematoma (General disorders) | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 4 | 7
Splenic infarction (Blood and lymphatic system disorders) | 2 | 0
Anaemia macrocytic (Blood and lymphatic system disorders) | 1 | 0
Anaemia of malignant disease (Blood and lymphatic system disorders) | 1 | 0
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 1 | 0
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0
Lymphadenitis (Blood and lymphatic system disorders) | 1 | 0
Spontaneous haematoma (Blood and lymphatic system disorders) | 1 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 4
Hypochromic anaemia (Blood and lymphatic system disorders) | 0 | 2
Anaemia haemolytic autoimmune (Blood and lymphatic system disorders) | 0 | 1
Anaemia of chronic disease (Blood and lymphatic system disorders) | 0 | 1
Pancytopenia (Blood and lymphatic system disorders) | 0 | 1
Cataract (Eye disorders) | 4 | 3
Glaucoma (Eye disorders) | 3 | 1
Open angle glaucoma (Eye disorders) | 1 | 1
Retinal detachment (Eye disorders) | 1 | 1
Maculopathy (Eye disorders) | 1 | 0
Ulcerative keratitis (Eye disorders) | 1 | 0
Blindness (Eye disorders) | 0 | 1
Endophthalmitis (Eye disorders) | 0 | 1
Myopia (Eye disorders) | 0 | 1
Ocular retrobulbar haemorrhage (Eye disorders) | 0 | 1
Optic ischaemic neuropathy (Eye disorders) | 0 | 1
Pterygium (Eye disorders) | 0 | 1
Uveitis (Eye disorders) | 0 | 1
Haematoma (Vascular disorders) | 3 | 3
Aortic aneurysm (Vascular disorders) | 1 | 1
Femoral arterial stenosis (Vascular disorders) | 1 | 1
Haemorrhage (Vascular disorders) | 1 | 1
Hypovolaemic shock (Vascular disorders) | 1 | 0
Angiodysplasia (Vascular disorders) | 0 | 1
Iliac artery embolism (Vascular disorders) | 0 | 1
Lymphoedema (Vascular disorders) | 0 | 1
Peripheral embolism (Vascular disorders) | 0 | 1
Thrombophlebitis (Vascular disorders) | 0 | 1
Varicose vein (Vascular disorders) | 0 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 2 | 0
Panniculitis (Skin and subcutaneous tissue disorders) | 1 | 0
Pemphigoid (Skin and subcutaneous tissue disorders) | 1 | 0
Photodermatosis (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 2
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 0 | 1
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 1
Depression (Psychiatric disorders) | 3 | 1
Mental status changes (Psychiatric disorders) | 1 | 3
Generalised anxiety disorder (Psychiatric disorders) | 1 | 0
Major depression (Psychiatric disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 2
Alcohol withdrawal syndrome (Psychiatric disorders) | 0 | 1
Alcoholism (Psychiatric disorders) | 0 | 1
Confusional state (Psychiatric disorders) | 0 | 1
Delirium tremens (Psychiatric disorders) | 0 | 1
Post-traumatic stress disorder (Psychiatric disorders) | 0 | 1
Suicide attempt (Psychiatric disorders) | 0 | 1
Hyperthyroidism (Endocrine disorders) | 2 | 0
Goitre (Endocrine disorders) | 1 | 1
Hypothyroidism (Endocrine disorders) | 1 | 0
Basedow's disease (Endocrine disorders) | 0 | 2
Adrenal disorder (Endocrine disorders) | 0 | 1
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 0 | 1
Ileostomy closure (Surgical and medical procedures) | 1 | 0
Shoulder arthroplasty (Surgical and medical procedures) | 1 | 0
Suprapubic catheter insertion (Surgical and medical procedures) | 1 | 0
Transurethral prostatectomy (Surgical and medical procedures) | 1 | 0
Hip arthroplasty (Surgical and medical procedures) | 0 | 3
Knee operation (Surgical and medical procedures) | 0 | 1
Pilonidal sinus repair (Surgical and medical procedures) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 2 | 4
Vertigo positional (Ear and labyrinth disorders) | 1 | 1
Hearing impaired (Ear and labyrinth disorders) | 0 | 1
Inner ear disorder (Ear and labyrinth disorders) | 0 | 1
Vestibular neuronitis (Ear and labyrinth disorders) | 0 | 1
Hypersensitivity (Immune system disorders) | 1 | 0
Sarcoidosis (Immune system disorders) | 0 | 1
Victim of crime (Social circumstances) | 1 | 0
Hydrocele (Congenital, familial and genetic disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dronedarone 400mg Bid (N=2291) | Placebo (N=2313)
Any Gastrointestinal disorders (Gastrointestinal disorders) | 573 | 478
Diarrhoea (Gastrointestinal disorders) | 222 | 142
Nausea (Gastrointestinal disorders) | 122 | 71
Any infections and infestations (Infections and infestations) | 508 | 533
Any general disorders and administration site conditions (General disorders) | 397 | 348
Oedema peripheral (General disorders) | 147 | 119
Fatigue (General disorders) | 115 | 90
Any musculoskeletal and connective tissue disorders (Musculoskeletal and connective tissue disorders) | 364 | 376
Any nervous system disorders (Nervous system disorders) | 362 | 365
Dizziness (Nervous system disorders) | 160 | 145
Any respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 315 | 318
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 120 | 96
Any investigation disorders (Investigations) | 298 | 199
Any cardiac disorders (Cardiac disorders) | 251 | 213
Any skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 235 | 174
Any injury, poisoning and procedural complications (Injury, poisoning and procedural complications) | 187 | 198
Any vascular disorders (Vascular disorders) | 179 | 187
Any metabolism and nutrition disorders (Metabolism and nutrition disorders) | 171 | 183
Any psychiatric disorders (Psychiatric disorders) | 106 | 125

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If no publication has occurred within 12 months of the completion of the study, the Investigator shall have the right to publish/present independently the results of the study. The Investigator shall provide the Sponsor with a copy of any such publication for comment at least 45 days before any submission for publication. If requested by the Sponsor, any submission shall be delayed up to 90 days, to allow the Sponsor to preserve its proprietary rights.